CLINICAL TRIAL: NCT03736980
Title: Beyond the Self and Back: Neuropharmacological Mechanisms Underlying the Dissolution of the Self
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 124
Record Dates: First submitted 2018-10-11; First posted 2018-11-09 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Four independent study groups
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Psilocybin Group 1 (Experimental): Group 1: randomized, placebo-controlled, double-blind, cross-over design
  Interventions: Drug: Placebo; Drug: Psilocybine
- Psilocybin Group 2 (Experimental): Group 2: randomized, placebo-controlled, double-blind, cross-over design
  Interventions: Drug: Placebo; Drug: Psilocybine
- Psilocybin Group 3 (Experimental): Group 3: randomized, placebo-controlled, double-blind, cross-over design
  Interventions: Drug: Placebo; Drug: Psilocybine
- Psilocybin Group 4 (Experimental): Group 4: randomized, placebo-controlled, double-blind, matched group design
  Interventions: Drug: Placebo; Drug: Psilocybine

INTERVENTIONS:
Drug: Placebo — 100% lactose
Drug: Psilocybine — Study Group 1: 0.250 mg/Kg weight Study Group 2: 0.200 mg/Kg body weight Study Group 3: 0.215 mg/Kg body weight Study Group 4: 0.315 mg/Kg body weight

SUMMARY:
The aim of the study is to identify neural signatures, behavioral and phenomenological expressions of self-related processes including: sense of agency, semantic distinction between self and other, selflessness (altruism), social agency, embodied self (interoception), perceptual functioning of dissolved self including hallucinations and crossmodal processing, and finally the mystical type dissolution of the self.

DETAILED DESCRIPTION:
Four placebo-controlled, double blind sets of procedures using psilocybin with four independent study groups will be conducted. The number of subjects, testing procedures and dose of psilocybin for each group are as follows: group 1 (20 subjects, EEG, questionnaires, 0.200 mg/Kg body weight), group 2 (30 subjects, functional magnetic resonance imaging (fMRI), questionnaires, 0.200 mg/Kg body weight), group 3 (10 subjects, fMRI, questionnaires, 0.215 mg/Kg body weight), study group 4 (80 subjects, blood serum and saliva parameters, questionnaires, fMRI (only in 20 subjects from this group), 0.315 mg/Kg body weight). The groups 1, 2 and 3 involve healthy volunteers. The group 4 involves healthy volunteer long-term and short-term meditators during a 5-day group meditation retreat. Together, 140 subjects will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers at the age of 20-40 y (Group 1, 2 and 3) and 20-60 y (Group 4)
* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained
* Willing to refrain from drinking alcohol the day before testing session, from drinking alcohol and caffeinated drinks at the testing days and from consuming psychoactive substances 2 weeks before testing days and for the duration of the study.
* Able and willing to comply with all study requirements
* Informed consent form was signed

Further inclusion criteria for the Study Group 4:

* over 5000 hours of meditation experience (40 participants)
* meditation naive (with no experience in meditation) or with a low experience in meditation (as a criterium the total amount of less than <100 hours of meditation experience will be used) (40 participants)

Exclusion Criteria:

* Poor knowledge of the German language
* Previous significant adverse response to a hallucinogenic drug
* Participation in another study where pharmaceutical compounds will be given
* Self or first-degree relatives with present or antecedent psychiatric disorders
* History of head trauma or fainting
* Recent cardiac or brain surgery
* Current use of medication known to affect brain function (e.g. benzodiazepines, antihistamines, aspirin, beta blockers, theophylline, azetazolamide, etc.)
* Concomitant therapy with potent inhibitors of cytochrome P-450 isoenzyme 3A4 (HIV protease inhibitors, macrolide antibiotics, azolederivative anti-infective agents)
* Presence of major internal or neurological disorders (including sepsis, pheochromocytoma, thyrotoxicosis, drug-induced fibrosis, familiar or basilar artery migraine)
* Cardiovascular disease (hypertonia, coronary artery disease, heart insufficiency, myocardial infarction within the past 6 months, coronary spastic angina)
* Peripheral vascular disease (thromboangiitis obliterans, luetic arteritis, severe arteriosclerosis, thrombophlebitis, Raynaud's disease)
* Liver or renal disease
* Pregnant or breastfeeding women (a urine pregnancy test will be done for all women capable of bearing children)
* Women of childbearing potential who are not using effective, established contraception, such as oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Further exclusion criteria for the Study Group 2, 3 and 4:

* Inability to lie still for about 60 minutes (e.g. because of sneezing, itching, tremor, pain)
* Metal parts in the body (piercings, brain aneurysm clip, implanted neural stimulator/cardiac pacemaker/defibrillator/Swan Ganz catheter/insulin pump, cochlear implant); metal shrapnel or bullet, ocular foreign body (e.g. metal shavings); current or previous job in metalworking industry
* Claustrophobia

The presence of any one of the above mentioned exclusion criteria will lead to exclusion of the subject.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
fMRI resting state activity (BOLD signal) | 60 minutes
EEG measurement (ERPs) | 60 minutes

SECONDARY OUTCOMES:
Subjective effects will be assessed with the 5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC) | 7 hours
  Total score of the 5D-ASC (5-Dimensional Altered States of Consciousness Rating Scale). Consists of 94 items which are rated on a visual analogue scale (100 millimeters in length). The scale ranges from 0 (no alterations) to 100 (maximum alterations). The items are scored by measuring the millimeters from the low end of the scale to the participant's mark (from 0 to 100).
Mood changes will be assessed with the Positive and Negative Affect Schedule (PANAS) | 7 hours
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of 10 positive and 10 negative valence word items. Each item is rated on a 5-point likert scale with a range from 1 (not at all) to 5 (very much). The final score of the PANAS Scale is the sum of the 10 terms on the positive scale in which a higher score indicates increased positive affect, with a subscale range of 10 to 50 and the sum of the 10 terms on the negative scale in which a higher score indicates more negative affect, with a subscale range of 10 to 50.

IPD SHARING:
Plan to Share IPD: No